CLINICAL TRIAL: NCT00220311
Title: A Multicenter Study to Confirm the Efficacy and Safety of Fludara i.v. (Fludarabine Phosphate, SH L 573), Administered in 6 Treatment Cycles (1 Treatment Cycle: 5-consecutive Day Dosing, Followed by an Observation Period of 23 Days) in Untreated Chronic Lymphocytic Leukemia Patients With Anemia and/or Thrombocytopenia
Brief Title: A Study to Confirm the Efficacy and Safety of Fludarabine Phosphate Administered in Untreated Chronic Lymphocytic Leukemia Patients With Anemia and/or Thrombocytopenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 303530; 90699
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Fludarabine Phosphate (Fludara)

INTERVENTIONS:
Drug: Fludarabine Phosphate (Fludara) — 6 cycles (1 cycle: 5 treatment days every 28 days)
  Other Names: BAY86-4864

SUMMARY:
The purpose of this study is to confirm the efficacy and safety of fludarabine phosphate administered with dose increasing in 6 cycles (1 cycle: 5 treatment days every 28 days) in untreated chronic lymphocytic leukemia (CLL) patients with anemia and/or thrombocytopenia.

DETAILED DESCRIPTION:
As of 29 May 2009, the clinical trial sponsor is Genzyme Corporation. NOTE: This study was originally posted by sponsor Schering AG, Germany, which was subsequently renamed to Bayer Schering Pharma AG, Germany.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed CLL
* Patients with hemoglobin concentration and/or platelet count below the institution's lower limit of normal
* Patients who have not received cancer chemotherapy or radiotherapy

Exclusion Criteria:

* Patients with apparent infections (including viral infections)
* Patients with serious complications (heart, liver, or kidney disease, etc.)
* Patients with a serious bleeding tendency (e.g., DIC)
* Patients with serious CNS symptoms
* Patients with fever >= 38°C (excluding tumor fever)
* Patients with interstitial pneumonia or pulmonary fibrosis
* Patients with active multiple cancers
* Patients receiving other investigational products within 6 months before registration in this study
* Patients with prior allergies to medications that are similar to the investigational product (purine nucleoside derivatives)
* Women who are pregnant, of childbearing potential, or lactating

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2000-11; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Response rate of final overall evaluation up to 6 treatment cycles (at about 6 months) | Up to 6 treatment cycles (at about 6 months)

SECONDARY OUTCOMES:
Response rate for measurable lesions / evaluable lesions / peripheral blood findings / bone marrow findings | Up to 6 treatment cycles (at about 6 months)
Duration of response and change of peripheral blood findings | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company